CLINICAL TRIAL: NCT06592092
Title: Clinical Study of QH104 Cell Injection for the Treatment of Meningeal Metastases of B7H3+ Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH10402-LMD-01
Record Dates: First submitted 2024-03-17; First posted 2024-09-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor; Meningeal Metastasis
Keywords: B7H3 positive；; CAR-γδT cell
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QH104 cell Injection(Allogenic B7H3 CAR-γδT cell) (Experimental): Plan to enroll 3 to 6 patients with meningeal metastasis of B7H3+ solid tumor with single or multiple local injections of allogenic B7H3 CAR-γδ T cells (3*107/ dose)
  Interventions: Biological: QH104 Cell injection

INTERVENTIONS:
Biological: QH104 Cell injection — Patients will first be pre-screened for B7H3 expression of tumor and exist Meningeal Metastases.

SUMMARY:
This is an open, single-arm, single-center, interventional clinical study. It is planned to enroll 3-6 patients with meningeal metastases from B7H3+ solid tumors and to explore, on a small scale, the efficacy of local injection of allogeneic B7H3 CAR-γδ T cells (3*107/dose) for the treatment of patients with meningeal metastases from B7H3+ solid tumors.

DETAILED DESCRIPTION:
This study is an open, single-arm, single-center, interventional clinical study. It is planned to enroll 3-6 patients with meningeal metastases from B7H3+ solid tumors and to explore, on a small scale, the clinical response to local injection of allogeneic B7H3 CAR-γδ T cells (3*107/dose) for the treatment of patients with meningeal metastases from B7H3+ solid tumors. During the period of cell therapy, the enrolled subjects may be given additional multiple infusions of cells, after imaging, neurological function, cerebrospinal fluid cytology or the investigator's assessment of the potential benefit of continuing cell therapy. It is recommended that the frequency of multiple infusions be 2 weeks each, and the interval between infusions can be adjusted at a later stage based on the PK and clinical symptoms of the subject after infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Have a histologically or cytologically confirmed solid malignant tumor with positive B7H3 expression;
3. ECOG ≤ 2 or KPS ≥ 60;
4. Life expectancy ≥ 8 weeks as assessed by the investigator;
5. Meningeal metastases (or with brain parenchymal metastases) from any solid malignancy that is refractory to standard treatment or for which no standard treatment is available and positive cerebrospinal fluid (CSF) cytology;
6. Substantially normal bone marrow reserve function and normal hepatic and renal function (laboratory tests are required to be satisfied prior to first treatment with QH104 Cell Injection):

   White blood cell count (WBC) ≥ 3 x 109/L; Lymphocyte count (LY) ≥ 0.8 x 109/L; Hemoglobin (Hb) ≥ 90 g/L; Platelet (PLT) ≥90×109/L; Albumin transaminase (ALT) & albumin transaminase (AST) < 1.5 x ULN; Serum creatinine (Cr) < 1.5 x ULN; Total bilirubin < 1.5 x ULN; PT & PTT ≤ 1.25 × ULN.
7. Pregnancy test should be negative for women of childbearing potential and both men and women agree to use effective contraception during treatment and for 1 year thereafter;
8. Be able to understand the requirements and matters of the trial and be willing to participate in the clinical study as required;
9. Sign the trial informed consent form.

Exclusion Criteria:

1. Targeted CNS irradiation within 7 days prior to receiving the first QH104 infusion;
2. Uncontrolled comorbidities including, but not limited to: persistent or active infections, symptomatic congestive heart failure, unstable angina, cardiac arrhythmias, or psychiatric/social conditions that would limit the patient's ability to comply with study requirements;
3. Has a known psychiatric or substance abuse disorder that would interfere with cooperation with trial requirements;
4. Is receiving treatment with any other investigational drug;
5. Have a confirmed diagnosis of an immunodeficiency disorder;
6. Have an active infection requiring systemic treatment;
7. Inability to perform an MRI;
8. Serious cardiovascular compromise: history of New York Heart Association (NYHA) class II or greater congestive heart failure, unstable angina, myocardial infarction or stroke within 6 months of first dose, or arrhythmia requiring treatment at screening;
9. Allergy to immunotherapy and related cells;
10. Prior treatment with CAR-T and other immune cell therapy;
11. Other reasons, in the opinion of the investigator, why participation in this study is not appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Clinical response | day14
  Evaluate the clinical response of QH104 cell injection in treating B7H3+ solid tumor meningeal metastases according to the Response Assessment in Neuro-Oncology (RANO) criteria

SECONDARY OUTCOMES:
Overall survival(OS) | 3month,6month,12month
  OS is defined as the time from QH104 cells infusion to the date of death.
Incidence of Adverse Events (AEs) | day14 and day 28
  AE is defined as any adverse medical event from the date of infusion to 14 days after QH104 infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versus host disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
quality of life(QoL) score | day 14 and day 28
  Use the M.D. Anderson Symptom Inventory for Brain Tumors (MDASI-BT) to evaluate quality of life for all enrolled subjects, with assessments conducted prior to each cell infusion and during follow-up.
Pharmacokinetic (PK) | At days 0, 1, 3, 7, and 14
  Assess the pharmacokinetics (PK) of QH104 cell infusion in B7H3+ solid tumor meningeal metastases by monitoring the quantity of CAR+ cells, their subpopulations following QH104 cell reinfusion.
Pharmacodynamic (PD) | At days 0, 1, 3, 7, and 14
  Assess the pharmacodynamics (PD) of QH104 cell infusion in B7H3+ solid tumor meningeal metastases by monitoring the quantity of CAR+ cells, their subpopulations, differentiation, exhaustion, and cytokine changes in the cerebrospinal fluid following QH104 cell reinfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China